CLINICAL TRIAL: NCT00294177
Title: Conformation of Beta Human Chorionic Gonadotropin During Chemotherapy for Persistent Gestational Trophoblastic Tumors Using Atomic Force Microscopy and Dual Polarisation Interferometry
Brief Title: Conformation of Beta Human Chorionic Gonadotropin During Chemotherapy for Choriocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9561702010; Taiwan NSC 94WFA0101857
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2006-02-20 (Estimated); Status verified 2006-02

CONDITIONS: Trophoblastic Neoplasms; Choriocarcinoma
Keywords: Trophoblastic Neoplasms; Chorionic Gonadotropin; Molecular Conformation
MeSH Terms: conditions — Trophoblastic Neoplasms; Choriocarcinoma | interventions — Microscopy, Atomic Force

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Device: atomic force microscopy
Device: dual polarisation interferometry

SUMMARY:
Gestational trophoblastic disease comprises a spectrum of diseases with different propensity for local invasion and metastasis, that is, partial and complete hydatidiform mole, choriocarcinoma, and placental site trophoblastic tumor.All trophoblastic tumors produce hCG, and monitoring of therapy is largely based on the determination of hCG in serum. The conformational change of tumor markers during antineoplastic chemotherapy for cancer and its clinical meaning has only been rarely studied. In this study, we will try to understand the conformational change of the tumor marker (hCG) during chemotherapy.

DETAILED DESCRIPTION:
The conformational change of human chorionic gonadotropin beta (hCG beta) during chemotherapy for gestational trophoblastic disease and its clinical meaning have not been well understood. In this study we will use atomic force microscopy and dual polarisation interferometry to measure the dimensions and conformational change of beta human chorionic gonadotropin during chemotherapy for persistent gestational trophoblastic tumors.

Gestational trophoblastic disease comprises a spectrum of diseases with different propensity for local invasion and metastasis, that is, partial and complete hydatidiform mole, choriocarcinoma, and placental site trophoblastic tumor. Persistent trophoblastic disease may develop both from partial and complete moles. All trophoblastic tumors produce human chorionic gonadotropin (hCG), and monitoring of therapy is largely based on the determination of hCG in serum. The more malignant forms also express excessive amounts of hCG beta, and simultaneous determination of hCG and hCG beta can be used to differentiate between molar disease and trophoblastic cancer, which is associated with a proportion of hCG beta exceeding 5%. Over glycosylated hCG has also been reported to be a characteristic of trophoblastic cancer, but its clinical utility remains to be established. The hCG beta level in serum is also used to evaluate prognosis with not only very high but also very low levels in relation to tumor burden being indicative of adverse prognosis. Because of that: 1). more malignant forms also express excessive amounts of hCG beta; 2). the half-life of hCG beta is longer than that of hCG; 3). the hCG beta /hCG ratio will increase when the levels decrease after successful therapy; and 4). the ratio has been found to increase during development of therapy-resistant disease, monitoring of gestational trophoblastic disease usually relies on human chorionic gonadotropin beta measurement. Treatment of choriocarcinoma is most often monitored by serial assay of hCG beta in serum until the levels are undetectable, and simultaneous determination of hCG beta can sometimes reveal a relapse earlier than hCG. Therefore, measurement of hCG beta is important in treatment of gestational trophoblastic tumors.

Human choriogonadotropin belongs to a family of heterodimeric glycoprotein hormones which are comprised of two noncovalently bonded subunits with four N-linked carbohydrates. During chemotherapy, the hCG beta molecules can be degraded. A study has been reported by crystallographic analysis by which they found that crystals of deglycosylated human chorionic gonadotropin has a hexagonal bipyramidal structure using a method of vapor diffusion against ammonium sulfate. Previously, conformation of the hCG molecule has rarely been studied. By chemical method, over glycosylated hCG has been reported to be a characteristic of trophoblastic cancer, but its clinical utility remains to be established. Photoelectric method is a newly developed method to study the conformation of the protein or glycoprotein molecules. As yet, there is no report about the conformation of hCG serial studies. Gestational trophoblastic tumor as well as other gynecological cancers often underwent antitumor chemotherapy and monitor by tumor markers. During the antineoplastic chemotherapies, the conformational change of tumor markers, including hCG beta in persistent gestational trophoblastic tumor for cancer and its clinical meaning has only been rarely studied. Up to the present time, it is still not well understood whether a conformational change or reduced stability of the heterodimer may occur during chemotherapy.

In this study we will use an atomic force microscopy (AFM) to probe the surface nanostructure of beta human chorionic gonadotropin. The conformational change of the beta human chorionic gonadotropin which is secreted by persistent gestational trophoblastic tumors during chemotherapy will be studied. We will also want to directly visualize a single molecular structure of beta human chorionic gonadotropin, and quantitative measurements of the dimensions of the glycoprotein will be provided. The average height calculated for each hCG beta particle will be measured and compared subsequently during chemotherapy. Moreover, a experiment using dual polarization interferometric (DPI) as a biosensor will also be performed, and the average monolayer thickness value will also be calculated. To investigate further the surface ultrastructure of a hCG beta molecule, a hCG beta sample at very low concentration will be scanned in vacuum by AFM. The higher-resolution images will clearly reveal the shape of hCG beta molecules. In addition, phase images of hCG beta molecules will be captured simultaneously with their height images, and the lateral dimensions of the shape of hCG beta molecules will then be measured and calculated. The average values calculated for the outside diameter and pore diameter will thus be obtained. This study will represent the first direct characterization of the surface ultrastructure of the hCG beta molecule at a nanometer scale. The physical measurements of the outer diameter, pore diameter, and protomer diameter in the hCG beta by AFM and DPI may suggest how to recognize hCG beta molecules, which constitute an important tumor marker during chemotherapy for persistent gestational trophoblastic tumors. Unraveling the molecular structure and measuring the dimensions of hCG beta may provide new directions for future application in clinical hCG beta sensor chips. In can also be likely that the dimensional change of hCG beta molecules may also have some clinical implications for persistent gestational trophoblastic tumors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of trophoblastic neoplasms
* Willing to be collected for the urine and 2 ml blood samples

Exclusion Criteria:

* Unwilling to be collected for the collect urine or 2ml blood sample

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2006-08; Study Completion 2008-07

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Jien Chen, Principal Investigator — Department or Obstetrics and Gynecology, National Taiwan university Hospital
Locations (1):
- National Taiwan University Hospital Department of Obstetrics and Gynecology, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Birken S, Armstrong EG, Kolks MA, Cole LA, Agosto GM, Krichevsky A, Vaitukaitis JL, Canfield RE. Structure of the human chorionic gonadotropin beta-subunit fragment from pregnancy urine. Endocrinology. 1988 Jul;123(1):572-83. doi: 10.1210/endo-123-1-572. PMID 2454811
- [Background] Swann MJ, Peel LL, Carrington S, Freeman NJ. Dual-polarization interferometry: an analytical technique to measure changes in protein structure in real time, to determine the stoichiometry of binding events, and to differentiate between specific and nonspecific interactions. Anal Biochem. 2004 Jun 15;329(2):190-8. doi: 10.1016/j.ab.2004.02.019. PMID 15158477
- [Background] Czajkowsky DM, Hotze EM, Shao Z, Tweten RK. Vertical collapse of a cytolysin prepore moves its transmembrane beta-hairpins to the membrane. EMBO J. 2004 Aug 18;23(16):3206-15. doi: 10.1038/sj.emboj.7600350. Epub 2004 Aug 5. PMID 15297878
- See also: library of National taiwan University Hospital — http://ntuml.mc.ntu.edu.tw